CLINICAL TRIAL: NCT07298226
Title: An Investigation Into the Immediate Effects of Atlanto-Occipital Joint Mobilization on Head Posture, Respiratory Function, and Cervical Range of Motion in Individuals With Forward Head Posture
Brief Title: Immediate Effects of Atlanto-Occipital Mobilization on Head Posture, Respiratory Function, and Neck Mobility in Forward Head Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Mesut Arslan, assistant professor, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BP-M
Record Dates: First submitted 2025-12-05; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Forward Head Posture
Keywords: Forward head posture; Atlanto-occipital joint mobilization; Cervical mobility; Respiratory function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Individuals included in the study will be allocated by block randomization into an intervention group (atlanto-occipital joint mobilization) and a control group (sham application).
Who Masked: Outcomes Assessor
Masking Description: The researcher performing the measurements will be blinded to the group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization group (Experimental): The intervention group will receive atlanto-occipital joint mobilization.
  Interventions: Other: Atlanto-occipital joint mobilization
- Sham group (Sham Comparator): The control group will receive the sham application.
  Interventions: Other: Sham application

INTERVENTIONS:
Other: Atlanto-occipital joint mobilization — The intervention group will receive a single session of atlanto-occipital joint mobilization.
  Arms: Mobilization group
Other: Sham application — The control group will receive a single session of sham intervention.
  Arms: Sham group

SUMMARY:
The purpose of this study is to investigate the immediate effects of atlanto-occipital joint mobilization on head posture, respiratory function, and cervical range of motion in healthy individuals with forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) is a common postural disorder characterized by the anterior displacement of the head relative to the shoulders. The estimated prevalence of FHP among individuals who use electronic devices frequently is reported to be high, affecting a significant portion of the general population. While postural correction exercises and ergonomic education are generally the first-line management strategies for FHP, manual therapy techniques (such as joint mobilizations and soft tissue therapy) are often recommended as an adjunct treatment. Additionally, various physiotherapy approaches, including stretching of the posterior cervical muscles, strengthening of the deep neck flexors, and respiratory exercises, can also be utilized. Specific mobilization of the atlanto-occipital joint is theorized to normalize arthrokinematics and reduce fascial restrictions in the suboccipital region. This is said to decrease neuromuscular tension, improve proprioceptive input, and restore optimal alignment, resulting in positive effects on head posture, cervical mobility, and respiratory function.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Being between the ages of 18 and 45.
* Having forward head posture according to craniovertebral angle measurement.

Exclusion Criteria:

* History of cervical surgery or trauma.
* Diagnosed cervical disc herniation or cervical stenosis.
* Presence of a diagnosed neurological and/or rheumatological disorder.
* Pregnancy.
* Presence of malignancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral Angle (CVA) for Forward Head Posture | Assessments will be performed at baseline (before the application) and immediately following the single-session intervention.
  Forward head posture will be assessed by measuring the craniovertebral angle (CVA) using a goniometer. The CVA is the angle between the horizontal line passing through the C7 spinous process and the line from the tragus of the ear to the C7 spinous process.
Respiratory Function assessed by Spirometry (FVC, FEV1, FEV1/FVC, PEF, FEF25-75%) | Assessments will be performed at baseline (before the application) and immediately following the single-session intervention.
  Respiratory function will be assessed using a spirometry device. The following parameters will be recorded and analyzed: Forced Vital Capacity (FVC), Forced Expiratory Volume in one second (FEV1), the FEV1/FVC ratio, Peak Expiratory Flow (PEF), and Forced Expiratory Flow at 25-75% of FVC (FEF25-75%).
Cervical mobility (Cervical Range of Motion (CROM)) assessed by Bubble Inclinometer | Assessments will be performed at baseline (before the application) and immediately following the single-session intervention.
  Cervical mobility (range of motion) will be assessed using a bubble inclinometer. Active range of motion will be measured in degrees for the movements of flexion, extension, lateral flexion (left/right), and rotation (left/right).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Rehabilitation, Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No